CLINICAL TRIAL: NCT00701506
Title: Patterned Electrical Neuromuscular Stimulation and Therapeutic Exercise for Osteoarthritis of the Knee: Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: RS Medical (Industry)
Collaborators: Accelerated Care Plus (Industry); Research Institute of Health and Science (RIHSE) (Unknown)
Responsible Party: William Carroll / Vice President of Reasearch and Product Development, RS Medical
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RSMED-OA-02
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Knee Osteoarthritis
Keywords: Knee; Osteoarthritis; Treatment; Electrostimulation
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 15 Patients (may be expanded) will receive stimulation with the following parameters:
  * 20-minute session, to each affected knee, 3 times per week for 12 weeks.
  * PENS for 20 minutes:
    * Tri-phasic Lower Extremity stimulation pattern based on activation timing of the quadriceps and hamstrings for strength training (50 Hz impulses for 200 ms every 1500 ms).
    * Minimal twitch for 5 minutes.
    * Moderate to strong, but well-tolerated twitch contractions for 15 minutes.
  * Electrodes placed on quadriceps and hamstrings.
  Interventions: Device: Patterned Electrical Neuromuscular Stimulation
- 2 (Placebo Comparator): 5 Patients (may be expanded) will receive stimulation with the following parameters:
  * 20-minute session, to each affected knee, 3 times per week for 12 weeks.
  * Placebo PENS for 20 minutes:
  * Electrodes placed on quadriceps and hamstrings.
  Interventions: Device: Placebo PENS

INTERVENTIONS:
Device: Patterned Electrical Neuromuscular Stimulation — * 20-minute session, to each affected knee, 3 times per week for 12 weeks.
  * PENS for 20 minutes:
    * Tri-phasic Lower Extremity stimulation pattern based on activation timing of the quadriceps and hamstrings for strength training (50 Hz impulses for 200 ms every 1500 ms).
    * Minimal twitch for 5 minutes.
    * Moderate to strong, but well-tolerated twitch contractions for 15 minutes.
  * Electrodes placed on quadriceps and hamstrings
  Other Names: The stimulator device is the Omnistim® FX² Pro Stimulation; Generator made by Accelerated Care Plus Corp (ACP).; The stimulator is used with Omnistim FX² Connector; Cables and ACP High Conductivity Electrodes.
  Arms: 1
Device: Placebo PENS — * 20-minute session, to each affected knee, 3 times per week for 12 weeks.
  * Placebo PENS for 20 minutes:
  * Electrodes placed on quadriceps and hamstrings.
  Other Names: The stimulator device is the Omnistim® FX² Pro Stimulation; Generator made by Accelerated Care Plus Corp (ACP).; The stimulator is used with Omnistim FX² Connector Cables; and ACP High Conductivity Electrodes.
  Arms: 2

SUMMARY:
The purpose of the study is to investigate the benefits of the Patterned Neuromuscular Electrical Stimulation (PENS) for the treatment of osteoarthritis. The rationale for this investigation is to assess the benefit of PENS in the alleviation of symptoms of osteoarthritis and elucidating the mechanism of action of PENS.

DETAILED DESCRIPTION:
There will be two study conditions; patients will be assigned to PENS treatment or to the control group.

Study arm 1 - 15 Patients (may be expanded) will receive stimulation with the following parameters:

* 20-minute session, to each affected knee, 3 times per week for 12 weeks.
* PENS for 20 minutes:

  * Tri-phasic Lower Extremity stimulation pattern based on activation timing of the quadriceps and hamstrings for strength training (50 Hz impulses for 200 ms every 1500 ms).
  * Minimal twitch for 5 minutes.
  * Moderate to strong, but well-tolerated twitch contractions for 15 minutes.
* Electrodes placed on quadriceps and hamstrings.

Study arm 2 - 5 Patients (may be expanded) will receive stimulation with the following parameters:

* 20-minute session, to each affected knee, 3 times per week for 12 weeks.
* Placebo PENS for 20 minutes:
* Electrodes placed on quadriceps and hamstrings.

A previous study was performed by the principal investigator to compare treatment of knee osteoarthritis with exercise vs a control group. The data from that study will be used to historically compare exercise with PENS treatment.

Primary Endpoints The following endpoints will be evaluated (between and within groups): Change in WOMAC osteoarthritis-specific status from baseline to end of treatment phase (12 weeks); Change in VAS.

Secondary Endpoints The following endpoints will be evaluated: Change in biochemical Synovial Fluid markers from baseline to end of treatment phase (12 weeks); MRI Data; Muscle strength; Change in pressure algometry of the knee joint; Change in patient self-reported and physician-reported global assessment from baseline to end of treatment (12 weeks); Change in pain intensity from baseline through the end of treatment phase (12 weeks); Change in physical function indices from baseline to end of treatment phase (12 weeks); Number of patients reporting 20% or more improvement in pain intensity; Number of patients recording 20% or more improvement in self-reported osteoarthritis overall questionnaire score; Number of patients indicating 20% or more improvement in self-reported and in physician-reported global assessment score.

Other Observations The following will also be monitored: Changes in prescription and over-the-counter medication usage (type used and amount taken); Adherence to treatment protocol (data from clinical treatment records); Safety of electrical stimulation and knee aspiration.

Primary Outcomes: Primary outcomes for this study is osteoarthritis-specific functioning, (WOMAC).

Osteoarthritis-specific functioning will be evaluated with the Western Ontario and McMaster Universities Osteoarthritis Index version 3.1 (WOMAC 3.1). The WOMAC 3.1 is a 24-item patient self-reported questionnaire assessing pain, stiffness, and physical function disability. The WOMAC is available in a Japanese version.

Pain intensity will be measured using a 10-centimeter visual analog scale (VAS scale). The scale will be anchored at one end with "0" and labeled "no pain at all," and at the other "10" and labeled "worst pain possible."

Secondary Outcomes: Secondary outcomes for this study are pain intensity, global assessment of function, physical functioning and safety.

Biochemical markers in knee joint fluid will be evaluated for change related to electrical stimulation. Synovial fluid will be aspirated, at baseline and after 12 weeks of electrical stimulation, from the osteoarthritic knee receiving stimulation. Fluid volume and acidity (i.e., pH), chondroitin 6-sulfate and chondroitin 4-sulfate concentrations, and hyaluronan (concentration, molecular weight and viscosity) will be assessed. Chondroitin sulfate isomers will be evaluated using high performance liquid chromatography. Hyaluronan viscosity will be determined using a capillary viscometer, molecular weight determined from viscosity, and concentration by protein assay.

MRI will be taken to evaluate the volume of the muscle group, thickness of the cartilage, and glucosaminoglycan content

Global assessment of function will be addressed with a single question; one for the patient and one for the treating physician. On a 10 cm visual analogue scale the following or similarly worded question will be rated: Considering all the ways OA has impacted your life {your patient's life} in the last month, how would you rate your {your patient's} condition today? The scale will be anchored at one end with "0" and the label "very poor," and at the other end with "10" and the label "very good."

Physical performance (objectively measured data) will be assessed using a timed up-and-go test. Quadriceps strength will be evaluated using a mechanical dynamometer.

Muscle strength should be conducted prior to the other physical performance measures to reduce bias due to fatigue. Responses to all questionnaires should be obtained prior to physical measurements, and then the physician should aspirate the treated knee.

Prescription medication regimen for the patients will be reported by the physician or study coordinator. The patient will report over-the-counter medication use.

Patient adherence to the stimulation protocol will be monitored through the clinical record.

Safety of electrostimulation and of the fluid aspiration procedure will be monitored via adverse events reports from the physician or study coordinator. Serious adverse events (i.e., fatal, life threatening, needing hospitalization) are not anticipated for electrostimulation or for aspiration of the knee. Anticipated adverse events for electrostimulation are minor (e.g., skin irritation), while for knee aspiration adverse events may include knee pain, swelling, stiffness, vasovagal or syncopal reaction.

ELIGIBILITY:
Inclusion Criteria:

* Patient may have evidence of osteoarthritis (radiographic and/or by patient symptoms report) in more than one joint, however, osteoarthritis of one knee has been the patient's primary complaint and the focus of treatment.
* Radiographic evidence, within 6 months of enrollment, of osteoarthritis of the knee receiving treatment.
* Kellgren and Lawrence osteoarthritis classification grade 1, 2 or 3 (i.e., indicative of cartilage still remaining in joint).
* Average rating of pain associated with osteoarthritis of knee greater than or equal to 4 cm (on a 10 cm visual analog scale).
* Stiffness in knee(s) lasts less than 30 minutes (to demonstrate that stiffness is not from a more serious condition)
* Agrees to follow their randomized treatment plan and use the device.
* At least 18 years old.
* Signed informed consent.
* Erythrocyte Sedimentation rate greater than 40 mm/hour (Higher rates may be indicative of RA)
* Agrees to follow the randomized treatment plan and use of the stimulation device.

Exclusion Criteria:

* Hypersensitivity to electrical stimulation.
* Undergone within 3 months of enrollment, corticosteroid or viscosupplementation (i.e., hyaluronate) injections to the effected knee.
* If taking medications such as oral steroids, non-steroidal anti-inflammatories, or acetaminophen, patient has been on a stable dose for at least 3 months prior to enrollment. (The criteria should match the prior retrospective data studies.)
* If taking chondroprotective supplements (e.g., glucosamine and chondroitin sulfate), patient has been on a stable dose for at least 3 months prior of enrollment.
* Pathologic process at the knee (congenital defect or blunt trauma leading to structural defect such as torn anterior cruciate or meniscus ligaments).
* Problems due to mechanical/anatomical deformities (i.e., valgus greater than 5 degrees or varus greater than 1.5 degrees)
* Women who are, or plan to become pregnant during the clinical investigation.
* Known malignancy or cancer.
* Morbid obesity (BMI > 40).
* Serious or uncontrolled systemic illness (e.g., autoimmune disease, rheumatoid arthritis, diabetes mellitus or renal failure).
* Implanted devices such as a cardiac pacemaker or defibrillator
* Concurrent use of another electrical stimulation device for treatment of knee symptoms.
* Ongoing enrollment, or discontinued enrollment within the last 30 days, in another clinical trial for medical devices or biologic agents.
* Relationship other than medical (e.g., spouse or employee of investigator) with principal investigator(s) and their staff which may bias patient reports.
* Relationship with another person enrolled in the clinical investigation.
* Unable to complete the study per the investigational plan or unable to complete the case report forms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-05; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Primary outcomes for this study are osteoarthritis-specific functioning, (WOMAC - Western Ontario and McMaster Universities Osteoarthritis Index version 3.1 in Japanese) and pain intensity measured with a VAS Scale (10-centimeter visual analog scale). | Baseline and weeks 4, 8, 12, 16, 20, 24

SECONDARY OUTCOMES:
Pain intensity, global assessment of function, physical performance, quad strength and safety. Knee joint synovial fluid will be aspirated and MRI imaging of the muscle/joint occurs at baseline and at week 12. Prescription/OTC medication reported. | Measurement timeframes discussed above or at baseline and weeks 4, 8, 12, 16, 20, 24

CONTACTS AND LOCATIONS:
Overall Officials: William Carroll, Study Director — RS Medical
Locations (1):
- Osaka General Medical Center, Osaka, Japan